CLINICAL TRIAL: NCT04072380
Title: A Phase 2, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of 2 mg and 4 mg SUVN-G3031 Compared to Placebo in Patients With Narcolepsy With and Without Cataplexy
Brief Title: A Study to Evaluate Safety, and Efficacy of SUVN-G3031 (Samelisant) in Patients With Narcolepsy With and Without Cataplexy
Acronym: SUVN-G3031
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suven Life Sciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTP2S13031H3
Expanded Access: NCT05530447 (No longer available)
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Narcolepsy
Keywords: SUVN-G3031; Narcolepsy with and without cataplexy; Cataplexy; Narcolepsy Type 1; Narcolepsy Type 2; Excessive Daytime Sleepiness (EDS); Histamine H3 receptor; Samelisant
MeSH Terms: conditions — Narcolepsy; Cataplexy; Disorders of Excessive Somnolence | interventions — samelisant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SUVN-G3031 2mg (Experimental): Orally taken once daily for 14 days
  Interventions: Drug: SUVN-G3031
- SUVN-G3031 4mg (Experimental): Orally taken once daily for 14 days
  Interventions: Drug: SUVN-G3031
- Placebo (Placebo Comparator): Orally taken once daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SUVN-G3031 — SUVN-G3031 Tablets
  Other Names: Samelisant
  Arms: SUVN-G3031 2mg; SUVN-G3031 4mg
Drug: Placebo — Placebo Tablets
  Arms: Placebo

SUMMARY:
This study is of an investigational drug called SUVN-G3031 (Samelisant) as a possible treatment for narcolepsy with cataplexy or narcolepsy without cataplexy. The main purpose of this study is to learn how well the study drug works and how safe the study drug is compared to placebo.

DETAILED DESCRIPTION:
This is a Phase 2, double-blind, placebo-controlled, parallel-group, multicenter study to evaluate the safety, tolerability, pharmacokinetics (PK), and efficacy of SUVN-G3031 compared to placebo in participants with narcolepsy with and without cataplexy. Participants will be randomized at a ratio of 1:1:1 to 2 mg SUVN-G3031, 4 mg SUVN-G3031, or placebo. Each participant will receive study drug once daily, in a tablet formulation, for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18 to 65 years (adult), inclusive.
* Have narcolepsy with or without cataplexy (Na-1 or Na-2) based on the International Classification of Sleep Disorders (3rd edition) criteria (new or previously diagnosed).
* Have undergone a multiple sleep latency test (MSLT) study showing an MSLT of ≤ 8 minutes.
* An Epworth Sleepiness Scale (ESS) score of ≥ 12; and mean Maintenance of Wakefulness Test (MWT) time of < 12 min.
* Body mass index ranging from 18 to < 45 kg/m2
* Negative urine drug screen.
* A woman must be either not of childbearing potential or of childbearing potential practicing highly effective methods of birth control.
* Willingness to complete the study protocol with full compliance with procedures and sign an informed consent form (ICF).

Exclusion Criteria:

* Habitual wake-up time after 8 AM as assessed by sleep diary, habitual sleep time of < 6 hours, and habitual bedtime past 1 AM as determined by sleep diary entries.
* Use of any investigational therapy within the 30-day period prior to enrollment.
* Excessive caffeine (defined as > 600 mg/per day) use at least 1 week prior to baseline assessments and during the course of the trial.
* Nicotine dependence that has an effect on sleep (eg, a patient who routinely awakens at night to smoke).
* Use of concurrent medications prescribed to treat narcolepsy as specified including stimulants, antidepressants and sodium oxybate.
* Current diagnosis of or past treatment for syndromes known to cause sleep disruption or any other cause of daytime sleepiness.
* Clinically significant ECG abnormalities.
* An occupation requiring variable shift work, night shifts, or frequent overnight travel which disrupts sleep patterns.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2019-09-21 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (39):
  - Sleep Disorders Center o f Alabama, Birmingham, Alabama
  - Santa Monica Clinical Trials, Los Angeles, California
  - Southern California Institute for Respiratory Diseases, Inc., Los Angeles, California
  - Pacific Research Network, Inc., San Diego, California
  - SDS Clinical Trials Inc., Santa Ana, California
  - Meris Clinical Research, Brandon, Florida
  - Teradan Clinical Trials, Brandon, Florida
  - St. Francis Medical Institute, Clearwater, Florida
  - PDS Research, Kissimmee, Florida
  - Sleep Medicine Specialists of South Florida, PA, Miami, Florida
  - Ivetmar Medical Group, LLC, Miami, Florida
  - Florida Pediatric Research Institute, Winter Park, Florida
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - NeuroTrials Research Inc, Atlanta, Georgia
  - The Neuro Center, Gainesville, Georgia
  - IACT Health, Lawrenceville, Georgia
  - Sleep Practitioners, LLC, Macon, Georgia
  - IACT Health, Rincon, Georgia
  - Clinical Research Institute, Stockbridge, Georgia
  - Helene A. Emsellem, MD PC, Chevy Chase, Maryland
  - Bronson Sleep Health, Portage, Michigan
  - Clinical Neurophysiology Services, Sterling Heights, Michigan
  - St Lukes Hospital, Sleep Medicine & Research Center, Chesterfield, Missouri
  - Clayton Sleep Institute, St Louis, Missouri
  - Research Carolina Elite, Denver, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Ohio Sleep Medicine Institute, Canton, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Intrepid Research, LLC, Cincinnati, Ohio
  - Cleveland Clinic, Sleep Disorders Center, Cleveland, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Respiratory Specialists, Wyomissing, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Bogan Sleep Consultants, Columbia, South Carolina
  - Lowcountry Lung Critical Care, North Charleston, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas
  - Roadrunner Research, San Antonio, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
- Canada (2):
  - Medical Arts Health Research Group, Kelowna, British Columbia
  - Jodha Tishon Inc, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nirogi R, Shinde A, Goyal VK, Ravula J, Benade V, Jetta S, Pandey SK, Subramanian R, Chowdary Palacharla VR, Mohammed AR, Abraham R, Dogiparti DK, Kalaikadhiban I, Jayarajan P, Jasti V, Bogan RK. Samelisant (SUVN-G3031), a histamine 3 receptor inverse agonist: Results from the phase 2 double-blind randomized placebo-controlled study for the treatment of excessive daytime sleepiness in adult patients with narcolepsy. Sleep Med. 2024 Dec;124:618-626. doi: 10.1016/j.sleep.2024.10.037. Epub 2024 Oct 30. PMID 39504585
- [Derived] Nirogi R, Mudigonda K, Bhyrapuneni G, Muddana NR, Shinde A, Goyal VK, Pandey SK, Mohammed AR, Ravula J, Jetta S, Palacharla VRC. Safety, Tolerability, and Pharmacokinetics of SUVN-G3031, a Novel Histamine-3 Receptor Inverse Agonist for the Treatment of Narcolepsy, in Healthy Human Subjects Following Single and Multiple Oral Doses. Clin Drug Investig. 2020 Jul;40(7):603-615. doi: 10.1007/s40261-020-00920-8. PMID 32399853

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SUVN-G3031 2mg | SUVN-G3031 4mg | Placebo
Started | 63 | 64 | 63
Safety Population | 63 | 63 | 62
Intent-to-treat (ITT) Population | 54 | 53 | 57
Completed | 51 | 50 | 53
Not Completed | 12 | 14 | 10
Not completed — Adverse Event | 4 | 6 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 1
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 2 | 3
Not completed — Intercurrent Illness and Others | 3 | 5 | 6

BASELINE CHARACTERISTICS:
Population: A total of 188 (98.9%) patients who were randomized to specific treatment sequence were included in the safety population and this population is considered for baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | SUVN-G3031 2mg | SUVN-G3031 4mg | Placebo | Total
Number analyzed (Participants) | 63 | 63 | 62 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (8.59) | 34.0 (10.0) | 33.6 (10.02) | 32.5 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 44 | 44 | 133
  Male | 18 | 19 | 18 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 11 | 6 | 21
  Not Hispanic or Latino | 59 | 52 | 56 | 167
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 3 | 7 | 2 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 13 | 16 | 14 | 43
  White | 47 | 38 | 43 | 128
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 3 | 4 | 13
  United States | 57 | 60 | 58 | 175
Epworth Sleepiness Scale (ESS) [Mean (Standard Deviation); unit: units on a scale] — The Epworth Sleepiness Scale (ESS) is a patient-reported questionnaire consisting of 8 questions. Each of the items are rated on a 4-point scale (0-3), based on the usual chances of dozing off or falling asleep while engaged in eight different activities. The total ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. Higher values represent a worse outcome.
  units on a scale | 17.3 (2.76) | 17.5 (2.84) | 17.1 (3.03) | 17.3 (2.86)
Clinical Global Impression of Severity (CGI-S) [Mean (Standard Deviation); unit: units on a scale] | 4.7 (0.80) | 4.8 (0.83) | 4.7 (0.87) | 4.8 (0.83)
Maintenance of Wakefulness Test (MWT) [Mean (Standard Deviation); unit: minutes] | 5.166 (4.466) | 6.141 (4.073) | 6.242 (4.158) | 5.846 (4.243)
Patient Global Impression of Change (PGI-C) [Mean (Standard Deviation); unit: units on a scale] | 4.8 (1.08) | 4.7 (1.03) | 4.8 (1.01) | 4.8 (1.04)

OUTCOME MEASURES:

1. Primary Outcome: Epworth Sleepiness Scale
Description: The Epworth Sleepiness Scale (ESS) is a patient-reported questionnaire consisting of 8 questions. Each of the items are rated on a 4-point scale (0-3), based on the usual chances of dozing off or falling asleep while engaged in eight different activities. The total ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. Higher values represent a worse outcome.
Time Frame: Change from baseline in the mean total ESS score at Day 14
Population: Intent to treat (ITT) population is considered for outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SUVN-G3031 2mg | SUVN-G3031 4mg | Placebo
Number analyzed (Participants) | 54 | 53 | 57
score on a scale | -5.1 (5.00) | -5.6 (5.46) | -3.3 (4.61)
Statistical Analysis 1: Comparison: SUVN-G3031 2mg vs SUVN-G3031 4mg vs Placebo; Test type: Superiority; p = 0.024, Mixed Models Analysis — Threshold for statistical significance was p≤0.05; Mixed model for repeated measures (MMRM)

2. Secondary Outcome: Clinical Global Impression of Severity
Description: The Clinical Global Impressions of Severity (CGI-S) scale is used to rate the severity of the patient's illness by clinician, on a 7-point scale with score ranging from 1 - 7. Higher values represent a worse outcome.
Time Frame: Change from baseline in the mean CGI-S score at Day 14
Population: Intent to treat (ITT) population is considered for outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SUVN-G3031 2mg | SUVN-G3031 4mg | Placebo
Number analyzed (Participants) | 54 | 52 | 55
score on a scale | -1.2 (1.24) | -1.4 (1.19) | -0.8 (1.17)
Statistical Analysis 1: Comparison: SUVN-G3031 2mg vs SUVN-G3031 4mg vs Placebo; Test type: Superiority; p = 0.009, Mixed Models Analysis — Threshold for statistical significance was p≤0.05; Mixed model for repeated measures (MMRM)

3. Secondary Outcome: Maintenance of Wakefulness Test
Description: Maintenance of Wakefulness Test (MWT) is an objective test of sleepiness that evaluates a person's ability to remain awake under soporific conditions for a defined period of time. In the MWT, time from start of the test to the time point of falling asleep will be measured, the total score can range from 0 - 30 minutes. Higher values represent a better outcome.
Time Frame: Change from baseline in the mean MWT score at Day 14
Population: Intent to treat (ITT) population is considered for outcome measure.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | SUVN-G3031 2mg | SUVN-G3031 4mg | Placebo
Number analyzed (Participants) | 54 | 52 | 57
minutes | 2.07 (4.68) | 4.25 (6.52) | 2.73 (7.00)
Statistical Analysis 1: Comparison: SUVN-G3031 2mg vs SUVN-G3031 4mg vs Placebo; Test type: Superiority; p = 0.734, Mixed Models Analysis — Threshold for statistical significance was p≤0.05; Mixed model for repeated measures (MMRM)

4. Other Pre Specified Outcome: Patient Global Impression of Change
Description: The PGI-C is based on a 7-point scale, where at each time point the patient will rate the change from baseline using the following query: "Since the start of the study, my overall status is: 1 = very much better; 2 = much better; 3 = a little better; 4 = no change; 5 = a little worse; 6 = much worse; 7 = very much worse." The PGI-C assessment will be based on change observed from baseline related to excessive daytime sleepiness rather than on the totality of the disease.
Time Frame: Analysis of Patient Global Impression of Change (PGI-C) at Day 14
Population: Intent to treat (ITT) population is considered for outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SUVN-G3031 2mg | SUVN-G3031 4mg | Placebo
Number analyzed (Participants) | 53 | 51 | 54
score on a scale | 3.2 (1.16) | 2.8 (1.10) | 3.7 (1.12)
Statistical Analysis 1: Comparison: SUVN-G3031 2mg vs SUVN-G3031 4mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis

5. Other Pre Specified Outcome: Clinical Global Impression of Change
Description: The CGI-C is based on a 7-point scale, where at each time point the physician will rate the change from baseline using the following query: "Compared to the patient's condition at admission to the project [prior to medication initiation], this patient's condition is: 1 = very much improved since the initiation of treatment; 2 = much improved; 3 = minimally improved; 4 = no change from baseline (the initiation of treatment); 5 = minimally worse; 6 = much worse; 7 = very much worse since the initiation of treatment." The CGI-C assessment will be based on change observed from baseline related to excessive daytime sleepiness rather than on the totality of the disease.
Time Frame: Analysis of Clinical Global Impression of Change (CGI-C) at Day 14
Population: Intent to treat (ITT) population is considered for outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SUVN-G3031 2mg | SUVN-G3031 4mg | Placebo
Number analyzed (Participants) | 54 | 53 | 57
score on a scale | 2.8 (1.01) | 2.6 (0.92) | 3.5 (0.91)
Statistical Analysis 1: Comparison: SUVN-G3031 2mg vs SUVN-G3031 4mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: From screening to Day 21
Arm/Group | SUVN-G3031 2mg | SUVN-G3031 4mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63 | 0/62
Other Adverse Events (participants affected / at risk) | 17/63 | 34/63 | 5/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SUVN-G3031 2mg (N=63) | SUVN-G3031 4mg (N=63) | Placebo (N=62)
Insomnia (Psychiatric disorders) | 6 (7) | 11 (11) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 3 (3) | 5 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 11 (13) | 2 (2)
Hot flush (Vascular disorders) | 3 (3) | 7 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT04072380/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT04072380/SAP_001.pdf